CLINICAL TRIAL: NCT06036004
Title: Oxytocin Substitution Therapy in Patients With AVP Deficiency (Central Diabetes Insipidus)
Brief Title: Oxytocin Substitution Therapy in Patients With Central Diabetes Insipidus
Acronym: OxyTUTION
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-01010; kt22ChristCrain
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Central Diabetes Insipidus (cDI)
Keywords: oxytocin (OXT); hypothalamic-pituitary axis; Arginine vasopressin (AVP); OXT deficiency; socio-emotional functioning; intranasal OXT
MeSH Terms: conditions — Diabetes Insipidus, Neurogenic; Diabetes Insipidus

STUDY DESIGN:
Intervention Model Description: double-blind randomised placebo-controlled trial: participants will be randomly assigned 1:1 to receive either treatment with intranasal OXT or intranasal placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study participants, study team (i.e., study nurses, study physicians, study psychologists), and further outcome assessors will be blinded after assignment to interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Product Intervention: intranasal OXT (Active Comparator): Intranasal OXT spray of 40 IU per ml (Syntocinon®).
  Interventions: Drug: Intranasal OXT
- Control Intervention: placebo nasal spray (Placebo Comparator): The placebo nasal spray will be identical in volume, labelling, container system, and other features.
  Interventions: Other: Placebo nasal spray

INTERVENTIONS:
Drug: Intranasal OXT — Syntocinon® contains the synthesized peptide OXT in a solution formulated to promote absorption through the nasal mucosa. Additional ingredients are E216 (propyl-4-hydroxybenzoate), E218 (methyl-4-hydroxybenzoate), and chlorobutanol hemihydrate. One bottle contains 5 ml, i.e., 200 IU of OXT in total. Each 0.1 ml nasal insulation delivers 4 IU of oxytocin.
  OXT (24 IU twice daily) is given for 28 (± 2) days of treatment.
  Arms: Study Product Intervention: intranasal OXT
Other: Placebo nasal spray — The placebo will contain no OXT but, otherwise, be identical to the intranasal OXT product with respect to the other ingredients.
  Placebo is given twice daily for 28 (± 2) days of treatment.
  Arms: Control Intervention: placebo nasal spray

SUMMARY:
This randomized, placebo-controlled, double-blind trial aims to investigate intranasal OXT as a novel therapeutical option in central diabetes insipidus (cDI) to improve psychological symptoms and socio-emotional functioning.

Optionally, patients can present for additional assessments in sub-studies:

* fMRI sub-study at day 14 (± 2 days) (one additional visit)
* Social-stress sub-study at day 14 (± 2 days) (one additional visit)

DETAILED DESCRIPTION:
Arginine vasopressin (AVP) and oxytocin (OXT) are hormones released into circulation from the posterior pituitary. While AVP acts mainly in the kidneys and causes reuptake of free water, OXT is well-known for its key role in the regulation of complex social-emotional functioning including attachment and pair bonding, fear possessing, emotion recognition, and empathy.

Disruption of the hypothalamic-pituitary axis can cause AVP deficiency

- known as central diabetes insipidus (cDI) - characterized by polyuria and polydipsia. Once diagnosed, desmopressin (an AVP receptor analogue) can be effectively used to treat diabetes insipidus. However, despite treatment with desmopressin, patients often report residual psychological symptoms, particularly heightened anxiety levels, depressed mood, impairment in social interactions, leading to an overall reduced quality of life.

Due to the anatomical proximity, local disruptions of the AVP system could also disturb the OXT system leading to an additional OXT deficiency. The additional OXT deficiency could explain (at least partially) the residual psychological deficits in patients with cDI. OXT replacement therapy to improve psychological symptoms would have great clinical implications. This randomized, placebo-controlled, double-blind trial aims to investigate intranasal OXT as a novel therapeutical option in cDI to improve psychological symptoms and socio-emotional functioning.

Optional fMRI sub-study: Participants will undergo a structural sequence to investigate grey and white matter anatomy (T1- weighted). Functional neuronal responses will be assessed through the surrogate of blood oxygenated level dependent (BOLD) signal, an indirect measure of neural activity. Three functional sequences (echo planar imaging, EPI) will investigate group differences in various aspects of brain activity: a resting state sequence and the EFMT.

Optional Social-stress sub-study: The three main components are an anticipation phase, a 5-minute interview, and a surprise mental arithmetic task. Acute stress is measured by cortisol increase.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a confirmed diagnosis of central diabetes insipidus based on accepted criteria
* Heightened anxiety levels (STAI - Trait subscale ≥ 39 score points) or alexithymia levels (impaired ability to identify and describe feelings; TAS-20 total ≥ 52 score points)
* Stable hormone replacement therapy for at least three months with desmopressin and, in case of additional anterior pituitary deficiencies, with the respective substitution therapies.

Exclusion Criteria:

* Participation in a trial with investigational drugs within 30 days
* Active substance use disorder within the last six months
* Consumption of alcoholic beverages >15 drinks/week
* Current or previous psychotic disorder (e.g., schizophrenia spectrum disorder)
* Pregnancy and breastfeeding within the last eight weeks
* Unwilling to use a medically acceptable form of contraception throughout the study period (female of childbearing potential only)
* Prolonged QTc-time >470 ms assessed with a 12-lead electrocardiogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in State-Trait Anxiety Inventory (STAI) questionnaire to assess general anxiety levels | Day 0, day 1, day 14, day 28
  Questionnaire with scores ranging from 1 ("almost never") to 4 ("almost always"). The STAI has two sub-scales, the State-Anxiety Scale (STAI-S; 20 items) and the Trait-Anxiety Scale (STAI-T; 20 items). The STAI-S evaluates the current state of anxiety, asking how respondents feel "right now," using items that measure subjective feelings of apprehension, tension, nervousness, worry, and activation/arousal of the autonomic nervous system. The STAI-T evaluates relatively stable aspects of "anxiety proneness," including general states of calmness, confidence, and security. The total scores range from 20 to 80, with higher scores indicating more pronounced anxiety. A score above 39/80 indicates clinically significant anxiety symptoms.
Change in EmBody/EmFace to assess recognition of facial and body expressions | Day 0, day 1, day 28
  The EmBody and EmFace subtasks comprise each of 42 stimuli showing body or facial expressions of angry, happy, or neutral affect. Stimuli last 1.5 seconds at 24 frames per second and are geometrically and optically standardised to prevent biases induced by ethnic cues. Each trial consists of one point-light display (PLD), followed by a response window during which participants are asked to indicate via mouse input which emotion they believe was portrayed in the PLD in a three-option forced-choice format (angry-neutral-happy). The total correct classification scores range from 0 to 42 (for each sub-task), with higher scores indicating more correct recognition of facial & body expressions.

SECONDARY OUTCOMES:
Change in Facial emotion recognition task (FERT) to assess emotion recognition and empathy | Day 0, day 28
  The FERT assesses the recognition of basic emotions. The task includes ten neutral faces and 160 faces that express one of four basic emotions (i.e., happiness, sadness, anger, and fear), with pictures morphed between 0% (i.e., neutral) and 100% in 10% steps. Stimuli are shown in random order for 500 ms, followed by the rating screen, where participants have to indicate the correct emotion. The outcome measure is accuracy (proportion correct).
Change in Multifaceted Empathy Test (MET) to assess the cognitive and emotional aspects of empathy | Day 0, day 1, day 28
  The computer-assisted test consists of 40 photographs that showed people in emotionally charged situations. To assess cognitive empathy, the participants are required to infer the mental state of the subject in each scene and indicate the correct mental state from a list of four responses. Cognitive empathy is the percentage of correct responses in the total responses. To measure emotional empathy, the subjects are asked to rate how much they feel for an individual in each scene (i.e., explicit emotional empathy) and how much they are aroused by each scene (i.e., implicit emotional empathy) on a 1-9 point scale.
Change in Hamilton Anxiety Rating Scale (HAM) to assess the severity of anxiety symptoms | Day 0, day 28
  The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). The physician/psychologist is instructed to assess the extent to which the patient displays the given criterion. Each item is independently scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56 (<17 indicates mild severity, 18-24 mild to moderate severity, and 25-30 moderate to severe).
Change in Toronto Alexithymia Scale 20 (TAS-20) to assess emotions experienced by oneself or others | Day 0, day 28
  The TAS 20 has a three- factor structure: difficulty identifying and describing feelings and externally oriented thinking. It includes 20 items with scores ranging from 1 (strongly disagree) to 5 (strongly agree). The total scores range from 20 to 100, with higher scores indicating worse alexithymia. A score of ≥61 indicates alexithymia (difficulty understanding one's emotions), a score of 52 to 60 indicates possible alexithymia, and a ≤51 non-alexithymia.
Change in Autism-Spectrum Quotient Test (AQ) to assess the expression of ASD traits in an individual by his or her subjective self-assessment | Day 0, day 28
  The AQ consists of 50 items, with four choices for each item from "definitely agree" to "definitely disagree" and a total score from 0 to 50. A score above the proposed cut-off of 29 highlights significant traits of autism
Change in Beck's Depression Inventory II (BDI-II) to assess depression | Day 0, day 28
  It uses 21 items ranked from 0 (symptom absent) to 3 (severe symptoms) to measure the severity of depression. The minimum score is 0, and the maximum score is 63. In non-clinical populations, scores above 20 indicate depression. In those diagnosed with depression, the score ≤16, mild mood disturbance; 17 to 20, borderline clinical depression, 21 to 30, moderate depression, and score ≥31, severe depression.

OTHER OUTCOMES:
Change in Close third-person assessment | Day 0, day 28
  A telephone interview with a close third individual can be conducted to provide a subjective assessment at the beginning and the end of the treatment phase. Assessment will be done by rating 10 socio-emotional items such as "closeness to others," "anxious behaviour daily life," "empathic feeling," etc., by using unidirectional 100-point or bidirectional -50/+50-point visual analogue scales.

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof. Dr. med., Principal Investigator — University Hospital Basel, Department of Endocrinology, Diabetes & Metabolism
Locations (2):
- Erasmus University Medical Center Rotterdam, Rotterdam, Netherlands
- University Hospital Basel, Department of Endocrinology, Diabetes & Metabolism, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results of this study will be made available upon reasonable request to the corresponding author, following publication of the primary results. Data will be shared with qualified researchers for purposes of academic, non-commercial research, subject to approval of a methodologically sound proposal and completion of a data-sharing agreement. Requests will be evaluated in accordance with applicable ethical approvals, data protection regulations, and institutional policies. Access will require approval and a signed data access agreement. The Department of Clinical Research (DKF), University of Basel, will act as an independent Data Access Committee and securely store the data at the time of publication. Requests for data reuse may be submitted via dkf.unibas.ch/contact.